CLINICAL TRIAL: NCT07382284
Title: Long-Term Survival After Left Ventricular Assist Device Support (LVAD) Implantation in Patients With End-Stage Heart Failure: A Prospective, Observational, Multi-Center Cohort Study
Brief Title: Long-Term Survival After LVAD Implantation in End-Stage Heart Failure
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: First Affiliated Hospital of Harbin Medical University (Other); The Affiliated Hospital of Yangzhou University (Unknown); Qianfoshan Hospital (Other); Xinhua Hospital of Ili Kazak Autonomous Prefecture (Unknown); Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-577-02
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: End-stage Heart Failure
MeSH Terms: interventions — Drug Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Myocardial tissue samples obtained from the left ventricular apex during LVAD implantation surgery, which are routinely removed as part of standard surgical care and would otherwise be discarded after pathological examination, will be retained. Peripheral blood samples obtained from routine clinical blood testing will also be retained for research analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Left Ventricular Assist Device (LVAD) implantation — Left ventricular assist device (LVAD) implantation performed as part of routine clinical care for patients with end-stage heart failure. This study is observational in nature and does not assign, alter, or mandate any intervention. The decision to implant an LVAD, the type of device used, perioperative management, and postoperative treatment are determined solely by the treating clinical team according to standard clinical practice.
  Other Names: Mechanical circulatory support implantation

SUMMARY:
This is a prospective, observational, multi-center cohort study designed to evaluate long-term survival and clinical outcomes in patients with end-stage heart failure undergoing left ventricular assist device (LVAD) implantation.

Patients receiving LVAD implantation as part of routine clinical care will be enrolled and followed for up to 3-5 years. During the study period, data will be collected on baseline characteristics, preoperative medical therapy, intraoperative surgical information, in-hospital course, and long-term postoperative medication use, as well as survival status, major clinical outcomes, LVAD-related complications, and hospital readmissions.

In addition, myocardial tissue samples will be obtained from the left ventricular apex during LVAD implantation surgery. These tissue samples are routinely removed as part of the standard surgical procedure and would otherwise be discarded after pathological examination. Peripheral blood samples will also be collected at predefined time points as part of routine clinical blood testing. No additional surgical procedures or invasive interventions are required for this study.

This study does not involve any experimental treatment or changes to standard medical care. All treatments and follow-up assessments are determined by the treating physicians according to routine clinical practice.

The purpose of this study is to improve understanding of long-term outcomes after LVAD implantation and to explore potential biological factors associated with prognosis in patients with end-stage heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥18 years
2. Diagnosis of end-stage heart failure refractory to optimal medical therapy
3. Scheduled to undergo left ventricular assist device (LVAD) implantation as part of routine clinical care
4. Able to provide written informed consent for participation and biospecimen collection
5. Willing and able to comply with study procedures and long-term follow-up
6. Availability of left ventricular apical myocardial tissue obtained during LVAD implantation surgery
7. Availability of peripheral blood samples collected during routine clinical care
8. Patients treated at participating study centers

Exclusion Criteria:

1. Age <18 years
2. Prior implantation of a durable mechanical circulatory support device
3. Concomitant heart transplantation at the time of index surgery
4. Congenital heart disease requiring complex surgical repair
5. Active systemic infection or sepsis at the time of LVAD implantation
6. Known active malignancy with a life expectancy <1 year
7. Severe non-cardiac comorbidities limiting expected survival to less than 1 year (e.g., advanced liver failure, end-stage renal disease not eligible for renal replacement therapy)
8. Inability or unwillingness to provide informed consent
9. Pregnancy or breastfeeding at the time of enrollment
10. Inadequate quantity or quality of myocardial tissue or peripheral blood samples for planned analyses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of adult patients with end-stage heart failure undergoing left ventricular assist device (LVAD) implantation as part of routine clinical care. Participants are primarily enrolled from Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School; The First Affiliated Hospital of Zhejiang University School of Medicine; and The First Affiliated Hospital of Harbin Medical University. A smaller number of patients are also enrolled from Jinan Central Hospital and the Affiliated Hospital of Yangzhou University. All participating centers are tertiary referral hospitals with established LVAD programs.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-07-17 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical response after LVAD implantation | During longitudinal follow-up up to 5 years after LVAD implantation
  Patients will be classified as responders or non-responders based on predefined criteria.

SECONDARY OUTCOMES:
Genetic and molecular correlates of clinical response after LVAD implantation | Assessed during follow-up up to 3-5 years after LVAD implantation
  Genetic and molecular analyses will be performed using myocardial tissue obtained from the left ventricular apex during LVAD implantation and peripheral blood samples collected during routine clinical care. Genome-wide association analyses and expression quantitative trait locus (eQTL) analyses will be conducted to explore associations between genetic variation, gene expression profiles, and long-term clinical response after LVAD implantation. These analyses are exploratory and aim to characterize the biological background underlying heterogeneity in myocardial recovery among patients with end-stage heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- +86 025 83106666, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data, including genetic and molecular data generated from myocardial tissue and peripheral blood samples, will not be shared at this time due to ethical, legal, and regulatory considerations. In particular, the collection and use of human genetic data are subject to national regulations, and data sharing decisions will be evaluated after completion of data collection and analysis to ensure compliance with applicable laws and institutional policies.

REFERENCES:
- [Result] Drakos SG, Badolia R, Makaju A, Kyriakopoulos CP, Wever-Pinzon O, Tracy CM, Bakhtina A, Bia R, Parnell T, Taleb I, Ramadurai DKA, Navankasattusas S, Dranow E, Hanff TC, Tseliou E, Shankar TS, Visker J, Hamouche R, Stauder EL, Caine WT, Alharethi R, Selzman CH, Franklin S. Distinct Transcriptomic and Proteomic Profile Specifies Patients Who Have Heart Failure With Potential of Myocardial Recovery on Mechanical Unloading and Circulatory Support. Circulation. 2023 Jan 31;147(5):409-424. doi: 10.1161/CIRCULATIONAHA.121.056600. Epub 2022 Nov 30. PMID 36448446